CLINICAL TRIAL: NCT02555033
Title: Effects of Simultaneous Balance and Resistance Training on Strength, Power and Balance in Older Adults: A Stratified and Randomised Trial
Brief Title: Effects of Simultaneous Balance and Resistance Training in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kassel (Other)
Collaborators: University of Potsdam (Other)
Responsible Party: Principal Investigator, Nils Eckardt, MEd, University of Kassel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFPS1415
Record Dates: First submitted 2015-09-08; First posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Muscle Weakness
Keywords: Instability resistance training; unstable surface; elderly people
MeSH Terms: conditions — Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- M-RT (Experimental): Machine-based resistance training. Exercising 'traditional' machine-based resistance training.
  Interventions: Other: Resistance training
- M-IRT (Experimental): Machine-based instability resistance training; a similar training program with exercise-machines, but with additional unstable devices placed between participant and exercise-machine or floor respectively.
  Interventions: Other: Instability resistance training
- F-IRT (Experimental): Free weight instability resistance training; conducted free-weight resistance training on unstable devices using dumbbells instead of exercise-machines.
  Interventions: Other: Instability resistance training

INTERVENTIONS:
Other: Resistance training — traditional resistance training
  Arms: M-RT
Other: Instability resistance training — training under unstable conditions
  Arms: F-IRT; M-IRT

SUMMARY:
Aging results in a gradual decline of physical abilities and consequently in functional impairments which increases the risk of falls in elderly people. It has been shown, that balance and resistance training can counteract the effects of aging. The aim of this study was to investigate effects of instability resistance training (IRT), combining balance and resistance training, on measures of muscle strength / power and balance for falls in healthy community-dwelling older adults. Therefore 75 elderly people, aged 65 - 80 years (Mage = 70.4; SD = 4.3 years) were assigned into three intervention groups: machine-based (M-RT), machine-based instability (M-IRT), free weight instability resistance training (F-IRT). All three groups exercised over 10-weeks with two training sessions per week. Assessment of muscle strength (e.g. maximal isometric leg extension strength), power (e.g. chair rise test) and balance (e.g. gait, functional reach test) was conducted before and after training.

Based on the principle of training specificity, it is assumed, that groups to improve better within their respective training modality. Thus, the investigators hypothesis that regarding measures of strength and power, M-RT performs better than M-IRT, performs better than F-IRT. As to measures of balance, we hypothesis that F-IRT performs better that M-IRT, performs better than M-RT.

DETAILED DESCRIPTION:
Background:

In the course of aging, physical abilities gradually decline. Even though the cause of falls is assumed to be multifactorial, loss in muscle strength and balance control seems to be the most crucial intrinsic risk factors for falls.

Several meta-analysis and reviews emphasise positive effects of resistance, balance and combined exercise interventions on measure of strength, power and balance performance and thus on intrinsic (i.e., person-related) risk factors for falls. Pure balance as well as pure resistance training have been effective in improving postural control (e.g., gait measures, leg extension strength) and reducing risk of falling in elderly people. Combined resistance and balance training describes in general a sequential or concurrent training program, where resistance and balance exercises are executed in a consecutive order within the same training session. These exercise interventions have shown positive effects as well. Merging resistance and balance training, executing both simultaneously has not been investigated in regard to fall prevention in elderly people yet.

In the past 15 years, research of simultaneous resistance and balance training, so called 'instability resistance training' (IRT), has been grown. IRT utilises unstable devices (Swiss balls, BOSU® balls, wobble boards, etc.) and an external load (e.g., weights). This training modality has shown to affect core and lower limb muscle activation positively, improving balance and further having comparable gains in measures of strength analogue to traditional resistance training. Kibele and Behm, for example, found superior improvements in the single leg hop following an IRT in healthy young adults. They concluded in line with the principle of training specificity, that IRT induced higher balance adaptions, which were prominent in the balance demanding singe leg hop. Further, Behm and Colado recommended IRT for elderly people and there are studies investigating effects of different kinds of IRT on older adults. Granacher and colleagues examined effects of core instability strength training (CIT) on measures of trunk muscle strength, spinal mobility, dynamic balance and functional mobility in older adults. They found meaningful improvements in measures of strength, balance and mobility in comparison to a control group. Another study, investigating effects of a swiss ball exercise program on older adults, found positive effects on measures of physical fitness and balance in comparison to a control group. Based on used exercises, these studies focused on strengthening the core and improving mainly balance abilities. In a slightly different approach to improve balance in older women, Chulvi-Medrano and colleagues utilized a lower-limb training program using a unstable T-Bow® device. The training group improved in measures of dynamic, static and overall balance, whereas the control group experienced a decline or no change in balance abilities. All three aforementioned studies utilised unstable devices but none incorporated additional loads within their training programs, hence the resistance component of IRT is limited to bodyweight. Hence, there is a lack of literature supporting evidence for feasibility and effectiveness of IRT incorporating additional load as resistance to improve measures of strength, power and balance in elderly people.

To the investigators knowledge, no study has been conducted yet, investigating effects of IRT with additional load as resistance on risk factors for falls for elderly people.

Measures:

Data was acquired in our biomechanics laboratory. Questionnaires were completed in separated rooms. All tests were conducted and explained, using standardised verbal instructions regarding the test procedure to maintain equal treatment for all participants. A single assessment lasted 90 min per participant.

Strength / power assessment:

Well established clinical and biomechanical tests were administered to measure primary outcomes in muscle strength and power. In accordance with the recommendations of Granacher et al. strength assessments were performed after balance assessments to reduce interfering effects of muscle fatigue. Further, strength and balance tests were administered in a random order within their respective block. One practice trial was provided for every test. Test procedures were conducted according to the recommendations of Gschwind et al. if not stated otherwise. Two test trials were executed using the mean for further statistical analysis. Except for maximal isometric leg extension strength and hand grip strength. There, the better value of two consecutive trials was used for statistical analysis. In between the trials, sufficient recovery periods were provided to reduce fatigue.

Maximal isometric leg extension strength (ILES) was examined with a cable pull device (Takei A5002, Fitness Monitors, Wrexham, England) with an upright body posture. Individual cable lengths were chosen to ensure a knee angle of approximately 135°. Participants were asked to start "pull[ing] initially with a moderate intensity and slowly increase the intensity to maximum exertion while keeping the upper body extended and upright" to prevent injuries. To ensure upright posture, participants were instructed to maintain contact between shoulder and wall and not lift their scapula while pulling. The test was repeated with at least one minute between measurements. The ILES showed excellent test-retest reliability (ICC = .98) for leg extension strength.

To measure handgrip strength a Takei hand dynamometer (Takei A5401, Fitness Monitors, Wrexham, England) was used. Participants stood upright with their arm aligned to the body and squeeze the device as hard as they could, using the dominant hand. The handle's width was adjusted to the participant's hand size. The intermediate phalanges had to be placed on the inner handle. The Takei handy dynamometer showed excellent test-retest reliability (ICC = .95).

In addition to isometric strength, power tests were conducted. Supplementary to the standard Chair Rise Test (CRT) on stable surface, test trials were recorded while standing on a foam pad (AIREX©) as well. Participants had to stand up and sit down five times as quickly as they could, without the aid of their arms. Therefore, arms had to be folded across the upper body. Time was measured by an ordinary stop watch to the nearest .01 second. After the countdown "ready-set-go", testing time was started and stopped when participants were sitting down for the fifth time. For the CRT high test-retest reliability has been shown (ICC = .89).

In addition, a stair climb power test was administered. This test has shown meaningful associations with mobility performance and strength measures. Ascent and descent times were recorded separately and power was calculated with the following formula: P =((M x D) x g )/t, where P = Power (Watt), M = Body mass (kg), D = Vertical distance covered (meters), t = Time (seconds) and g = 9.8 (constant of gravity). Participants were instructed to walk quickly but safely up and down a 9-step flight of stairs (17 cm step height). Time was started after the cue to go and stopped when the second foot reached the top step and/or the floor, respectively. Use of the handrail was allowed for safety reasons. Time was measured with an ordinary stop watch to the nearest .01 second. Test-retest reliability has shown to be excellent (r = .99).

Balance:

Dynamic steady-state balance was tested while walking on a 10-m walkway, measuring temporal-spatial gait variables (stride length (cm), double support time (%), speed (m/s), step width (cm)) using a two-dimensional OptoGait© system (Microgait, Bozano, Italy). In addition the coefficient of variation was computed (CV = (SD/mean) x 100). The OptoGait© system showed high interclass correlation coefficients (ICC's = .93 - .99) and high concurrent validity between the OptoGait© system and a previously validated system. Participants were asked to walk for 10 m with their own footwear at a self-selected pace three times to calculate test-retest reliability. Because the OptoGait© system is able to record automatically, a starting signal was not necessary. A three-minute interval was given between individual trials to rest, save the data as well as to prepare for the next trial. At the start and the end of the walkway sufficient distance was provided to accelerate and decelerate safely. In addition, the first and last step was excluded from analysis to eliminate possible acceleration and deceleration bias. Each trial was recorded with 1000 Hz using the manufacture provided OptoGait© software running on a laptop computer (Lenovo ThinkPad T530).

Proactive balance was tested using the Functional Reach Test (FRT) and the Timed up and Go Test (TUG). The FRT measures the maximal distance participants were able to reach forward while standing. For this purpose, participants were instructed lift their dominant arm and to reach forward as far as they could without taking a step forward. Maximal reach distance (cm) was assessed. The FRT showed excellent test-retest reliability with elderly people (ICC = .92). FRT trials were repeated when participants were not able to maintain both feet on the ground at a fixed position. In addition to the standard FRT on solid surface, test trials were recorded while standing on a foam pad (AIREX©) as well. For the TUG, participants were asked to rise from a chair and walk three meters in their normal walking speed around a cone, return and sit down. Time for the TUG was recorded with an ordinary stopwatch to the nearest .01 second on the command "ready-set-go" and stopped as soon as the participants sat down. The TUG showed excellent test-retest reliability (ICC = .99) in older adults.

To test reactive balance, the Push and Release Test (PRT) was used. The PRT rates the postural response to a sudden perturbation. Participants were instructed to push backwards against the examiner's hands and to regain their balance after the examiner releases his hands. The number of steps required to regain balance was counted and the corresponding score was recorded (0 = 1 step, 1 = 2-3 small steps backwards with independent recovery, 2 = ≥4 steps with independent recovery, 3 = steps with assistance for recovery, 4 = fall or unable to stand without assistance). For a detailed description of the PRT see Jacobs and colleagues. The PRT showed high test-retest reliability (ICC = .84) with a sensitivity of 89% and a specificity of 85%.

Questionnaires:

Psychosocial functions were assessed using several questionnaires. Global cognition was tested using the MMSE, which is a reliable test for assessing cognitive function showing high test-retest reliability (r = .89). The CDT and FAB-D were used to assess executive function. Inter-rater reliability of the CDT was shown to be high (IRR = .92) with sensitivity and specificity values of .50 and .84, respectively. Falls self-efficacy was measured using the German version of the FES-I. This test has shown excellent internal validity (Cronbach's alpha = .96) and test-retest reliability (r = .96) to assess the level of fear of falling. To assess health-related physical activity, exercise and the amount of energy expenditure, FQoPA was conducted. Frey and colleagues showed that FQoPA score correlates with maximum oxygen uptake, indicating high validity (r = .42).

Design of the exercise intervention:

Participants were stratified into three intervention groups based on equal distribution of age and equal gender ratio. The allocation of the training program occurred randomly. Intervention group one conducted a 'traditional' machine-based resistance training (M-RT). Intervention group two (machine-based instability resistance - M-IRT) followed a similar training program with exercise-machines, but with additional unstable devices placed between participant and exercise-machine or floor respectively. The third intervention group conducted free-weight resistance training on unstable devices (F-IRT) using dumbbells instead of exercise-machines. All intervention groups trained for 10 weeks, twice per week on non-consecutive days for 60 min. The 10-week intervention period consisted of one week introductory phase and three major training blocks lasting three weeks each. Training intensity was progressively and individually increased over the 10-week training program by modulating load and sets for all groups and level of instability for group M-IRT and F-IRT. After week one, four and seven the training load (weight) was increased following 1RM (one repetition maximum - maximum amount of force that can be generated within one repetition) testing for each exercise. Since the load of 1RM is too heavy for untrained elderly, training load was calculated using the prediction equation provided by Epley, showing .03% deviation of actual achieved 1RM in squats with a correlation of .97. Instructors made sure that repetitions did not exceed 15-20, because 1RM predication accuracy is higher with fewer repetitions. Training under unstable conditions, especially with additional weight, implies a certain degree of accident risk. Therefore all instability exercises were secured by instructors and additional aids like boxes. Training has been supervised by skilled instructors. For the first two weeks the participant to instructor ratio was 5:1, afterwards 10:1.

Since effectiveness of resistance training to prevent falls has been reported frequently, intervention group one (M-RT) acted as an active control group. In a study by Orr and colleagues, participants with comparable baseline characteristics showed significant higher treatment effects in comparison to a passive control group (p < .001). Since the aim of the study was to compare an untested intervention (IRT) and an effective treatment (RT), the investigators decided to implement an active instead of a passive control group design.

Intervention program:

All three intervention groups conducted a resistance training program consisting of three main exercises, a warm-up and cool-down phase. Participants performed 10 min low-intensity stepping on a stair-walker as a brief warm-up in the beginning of each training session. The core part of the intervention exercises focused on strengthening leg extension muscles. Therefore squat-movements were chosen, as recommended by Flanagan and colleagues. M-RT and M-IRT groups performed squats on a Smith machine, fixing the barbell at hip level. Pilot testing revealed that shoulder and lower back mobility of elderly were too limited for fixing the barbell on the shoulders. In addition, the M-IRT group used instability devices (e.g. BOSU balls, wobble boards, inflatable discs) placed under the feet. Instability devices were used in the F-IRT group as well, but they performed the squat with dumbbells instead of a barbell. As a secondary leg extension exercise, leg-press for the M-RT and M-IRT (using instability devices put between feet and foot plate) were chosen. The front lunge (with dumbbells) was used as a secondary exercise by the F-IRT group. To strengthen the core, the bridge exercise was incorporated into the training program. Again, group M-IRT and F-IRT used instability devices placed under the shoulder and the feet in addition.

Statistics:

An a priori power analysis using G*Power 3.1 with an assumed type I error of .05 and a type II error of .10 (90% statistical power) was computed to determine an appropriate sample size to achieve statistically significant interaction effects. The calculations were based on a study assessing the effects core instability strength training in older adults. The analysis revealed the necessity of 54 participants (18 per group) to obtain medium (.24 ≤ f ≤ .39) "time x group" interaction effects. Considering the likelihood of dropouts we decided to recruit more than 66 participants to compensate a possible dropout rate of 20%.

Prior to main analysis normal distribution was tested with the Kolmogorov-Smirnov tests for each dependent variable. In addition, Levene's test for equality of variance was conducted. We tested baseline differences between groups with a one-way ANOVA or a Kruskal-Wallis test depending on distribution and homogeneity. In order to test the hypothesis, a 3 (group: M-RT, M-IRT & F-IRT) x 2 (time: pre- and post-test) ANOVA, with repeated measures on time was calculated. In case of distribution or homogeneity violations non-parametric Friedman and Kruskal-Wallis tests were computed to control results of parametrical tests and for non-parametrical variables. If differences were detected, non-parametrical results were expressed. Because Bonferroni-correction for multiple comparisons has been found too conservative, Ryan-Holm-Bonferroni adjusted post-hoc tests were used to analyse significant "time x group" interactions or tendencies (.051 ≤ p < .10). Independent t-tests or Mann Whitney-U were used to identify differences between groups. Ryan-Holm-Bonferroni corrected p-values were reported. In addition, differences in absolute training intensity within the last training block were analysed. Thus, the training load of the squat movements, which was common to all groups, was used. Differences were computed using a one-way ANOVA. Dependent on distribution and homogeneity, Ryan-Holm-Bonferroni adjusted post-hoc tests (independent t-test or Mann Whitney-U) were computed to detect differences between groups. Changes for all variables within groups were calculated by the formula ∆% = ((Meanpre / Meanpost) - 1) x 100. The effect size for ANOVAs' was determined by calculating Cohen's f. Following Cohen, f-values ≤ .24 indicate small effects, .25 ≤ f ≤ .39 indicate medium effects and f ≥ .40 indicate large effects. For post-hoc tests Cohen's d was calculated. Following Cohen, d-values ≤ .49 indicate small effects, .50 ≤ d ≤ .79 indicate medium effects and d ≥ .80 indicate large effects. Significance level was set at α = 5%. All analyses were performed using SPSS version 21.0 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* ability to walk independently without any gait aid

Exclusion Criteria:

* pathological ratings of the Clock Drawing Test (CDT),
* Mini-Mental-State-Examination (MMSE, < 24 points),
* Falls Efficacy Scale - International (FES-I, > 24 points),
* Geriatric Depression Scale (GDS, > 9 points),
* Freiburg Questionnaire of Physical Activity (FQoPA, < 1hour)
* Frontal Assessment Battery (FAB-D, < 18 points)
* any neurological, musculoskeletal or heart-related disease

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Maximal isometric leg extension strength (ILES) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in isometric strength, measured in N

SECONDARY OUTCOMES:
Fall self-efficacy Questionnaire | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in anxiety score
Dynamic Balance (stride velocity) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in stride velocity (m/s)
Dynamic Balance (stride length & step width) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in stride length and width (cm)
Dynamic Balance (double support) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in double support time (% of the stride cycle)
Proactivec Balance (timed up and go test) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in leg strength and procative balance (seconds)
Proactivec Balance (functional reach test) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in proactive balance (cm)
Reactive balance (push and release) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in reactive balance (score)
Power tests (chair rise test) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in muscle power (seconds)
Power tests (stair power test) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in muscle power (seconds)
Power tests (stair power test) | Pre test -> Intervention (10 weeks) -> Post test (within 2-5 days after the intervention)
  change in muscle power (watt)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Kibele, Prof., PhD, Study Chair — University of Kassel
Locations (1):
- University of Kassel, Kassel, Hesse, Germany

REFERENCES:
- [Result] Gschwind YJ, Kressig RW, Lacroix A, Muehlbauer T, Pfenninger B, Granacher U. A best practice fall prevention exercise program to improve balance, strength / power, and psychosocial health in older adults: study protocol for a randomized controlled trial. BMC Geriatr. 2013 Oct 9;13:105. doi: 10.1186/1471-2318-13-105. PMID 24106864
- [Result] Behm D, Colado JC. The effectiveness of resistance training using unstable surfaces and devices for rehabilitation. Int J Sports Phys Ther. 2012 Apr;7(2):226-41. PMID 22530196
- [Derived] Eckardt N. Lower-extremity resistance training on unstable surfaces improves proxies of muscle strength, power and balance in healthy older adults: a randomised control trial. BMC Geriatr. 2016 Nov 24;16(1):191. doi: 10.1186/s12877-016-0366-3. PMID 27881086